CLINICAL TRIAL: NCT04111276
Title: In Vivo Three-Dimensional Determination of Osteoarthritis Brace Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: BREG, Inc (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB20191576
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects diagnosed with osteoarthritis of the knee (Experimental): Subjects must be diagnosed with marked unicompartimental degenerative joint space narrowing.
  Interventions: Device: Breg Osteoarthritis Brace gait fluoroscopy; Other: Gait fluoroscopy without brace; Diagnostic Test: JointVue ultrasound; Diagnostic Test: Computer Tomography

INTERVENTIONS:
Device: Breg Osteoarthritis Brace gait fluoroscopy — Gait under fluoroscopy surveillance with brace
Other: Gait fluoroscopy without brace — Gait under fluoroscopy surveillance without brace
Diagnostic Test: JointVue ultrasound — JointVue ultrasound procedure to reconstruct 3D femoral and tibial bones
Diagnostic Test: Computer Tomography — Computer Tomography scan limited to the study knee and will image 6 inches distal on the tibia and 6 inches proximal on the femur

SUMMARY:
In vivo knee kinematics will be assessed for 20 subjects that have been clinically diagnosed with substantial unicompartmental osteoarthritis (OA) by one of the surgeons of Colorado Joint Replacement; this is the location from which participants will be recruited. The objective of this study will be to analyze subjects with symptomatic unicompartmental osteoarthritis under in vivo dynamic, weight-bearing conditions using video fluoroscopy to determine if present-day OA knee braces provide separation of the femoral condyle from the tibial plateau, thus avoiding excessive loads on the degenerative compartment.

DETAILED DESCRIPTION:
In vivo knee kinematics will be assessed for 20 subjects that have been clinically diagnosed with substantial unicompartmental osteoarthritis (OA) by one of the surgeons of Colorado Joint Replacement; this is the location from which participants will be recruited.

Enrollment will be increased to 24 subjects to account for any dropouts. Medial joint space narrowing will be clinically assessed in all patients on standing anteroposterior radiographs. The objective of this study will be to analyze subjects with symptomatic unicompartmental osteoarthritis under in vivo dynamic, weight-bearing conditions using video fluoroscopy to determine if present-day OA knee braces provide separation of the femoral condyle from the tibial plateau, thus avoiding excessive loads on the degenerative compartment.

Subjects will be asked to perform gait without the assistance of an offloading brace while under fluoroscopic evaluation. Then, each subject will be fitted with a Breg, off-the-shelf OA brace and will perform normal gait while under fluoroscopic surveillance. To ensure each brace was fitted properly, Breg will be asked to send either a sales representative or an engineer to the evaluation site. Therefore, the sales representative or engineer will be asked to fit their brace on each of the subjects.

Since the skeletal geometry is different for every person, computer aided design (CAD) models of the femur and tibia will be created for each specific subject. In order to create these CAD models, each subject will be asked to undergo a three-dimensional (3D) ultrasound using the JointVue proprietary software to reconstruct 3D femoral and tibial bones. A representative from JointVue will be present during data collection to conduct the ultrasound procedure in order to create the CAD models.

Participants will be asked to schedule a CT scan at Porter Adventist Hospital at their convenience to aid in the development of the bone models. To ensure subject safety, CT will be limited to the affected knee and the rest of patient's body will be protected from radiation with lead protection. The CT scan will be limited to the study knee and will image 6 inches distal on the tibia and 6 inches proximal on the femur.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient of Colorado Joint Replacement.
* Must be diagnosed with marked unicompartimental degenerative joint space narrowing.
* Bilateral subjects may not be included in the subject population

Exclusion Criteria:

* Pregnant, potentially pregnant or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study.
* Subjects who are unable to perform normal walking.
* Subjects who are unwilling to sign Informed Consent/ HIPAA documents.
* Does not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Komistek, PhD, Principal Investigator — University of Tennessee
Locations (3):
- United States (3):
  - Colorado Joint Replacement, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Diagnosed With Osteoarthritis of the Knee
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Diagnosed With Osteoarthritis of the Knee
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Medial Condylar Separation With Brace
Description: Medial condylar separation during gait
Time Frame: One day
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects Diagnosed With Osteoarthritis of the Knee
Number analyzed (Participants) | 20
mm | 0.60 (1.14)

2. Primary Outcome: Medial Condylar Separation Without Brace
Description: Medial condylar separation during gait
Time Frame: One day
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects Diagnosed With Osteoarthritis of the Knee
Number analyzed (Participants) | 20
mm | -1.05 (1.00)

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Subjects Diagnosed With Osteoarthritis of the Knee
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04111276/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04111276/SAP_001.pdf